CLINICAL TRIAL: NCT01920763
Title: Clinical Outcomes Following Parafascicular Surgical Evaluation of Intracerebral Hemorrhage: A Pilot Study
Brief Title: Observational Study of Safety and Outcomes After Minimally Invasive Surgery for Intracerebral Hemorrhage
Acronym: MiSPACE
Status: Withdrawn | Type: Observational
Why Stopped: Lack of recruitment.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MiSPACECan-001
Record Dates: First submitted 2013-07-22; First posted 2013-08-12 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2013-08

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Surgical evacuation; Minimally-invasive surgery
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical Patients: Patients with intracerebral hemorrhage who have been offered a parafascicular, minimally-invasive procedure for hematoma drainage, by the treating neurosurgeon.
  Interventions: Other: Clinical Measurement

INTERVENTIONS:
Other: Clinical Measurement — No direct interventions; study is observational and clinical assessments only will be performed.

SUMMARY:
This pilot study will examine the safety and the clinical outcomes after minimally invasive surgery (using a parafascicular technique guided by diffusion-tensor imaging) for intracerebral hemorrhage in patients selected according to evidence-based criteria. The investigators will compare 30 day and 90 day outcomes of patients who have surgery to that predicted by previously reported models for recovery after ICH, and will also describe any surgical complications related to the procedure.

The investigators hypothesize that this technique will have the same mortality rate and function outcome, if not better, when compared to the outcomes predicted by previous models.

DETAILED DESCRIPTION:
1.1 Intracerebral hemorrhage (ICH) morbidity, mortality, and functional outcomes. ICH is the most severe form of stroke: 30-day mortality is 40%, and 80% of survivors are physically disabled. Baseline hematoma volume and expansion are the most important determinants of outcome and are often therapeutic targets for trials. To date, there is no accepted medical therapy for ICH, particularly in supratentorial hematomas. Attempts to mitigate neuronal injury with treatments such as aggressive blood pressure lowering, hemostatic agents, reversal of anticoagulation, and surgical evacuation have been unsuccessful. We need an innovative approach to treat this lethal and disabling disease.

1.2 ICH surgery as a therapeutic approach. Mechanical and toxic effects of an accumulating intracerebral hematoma play an important pathophysiological role in ICH related brain injury. However, randomized controlled trials of hematoma evacuation have yielded inconsistent results. The largest randomized controlled trial of surgery for ICH failed to show a clinical benefit, possibly due to differences in surgical protocols, a 25% cross-over rate from medical to surgical arms, and substantial delays in onset-to-surgery times (median 3 days). This trial also raised the possibility that collateral injury to normal tissue during surgery can adversely affect outcome, as patients who appeared to benefit most were those with superficial and easily accessible hematomas. A subsequent meta-analysis indicated surgery may be beneficial for acute ICH with careful patient selection and short onset-to-surgery times. But at present, the surgical evacuation of ICH remains an unproven therapy.

1.3 Minimally invasive surgery for ICH. Traditionally, two of the strongest influences on treatment selection have been hematoma depth and dominance of the hemisphere involved, with a non-operative approach favoured for deep and dominant hematomas. In conventional clot evacuation, brain retraction is often required to maintain access to the lesion. Brain contusion and tissue injury is estimated to occur in 5-10% of cases after retraction, and can result in clinical deficits. Procedure related damage to the subcortical white matter has also been suggested to contribute to neurocognitive and affective changes after ICH evacuation. Minimally invasive surgery (MIS) offers potential advantages over conventional craniotomy, and several groups have developed and examined such techniques. Again, results have been conflicting and improved functional outcome has not been consistently demonstrated. MIS techniques specifically designed to avoid eloquent cortex and subcortical tracts during hematoma evacuation present a new and exciting paradigm for ICH therapy

1.4 Diffusion tensor imaging (DTI) and parafascicular surgical evacuation of ICH. Cerebral white matter is organized into well-defined fascicles and tracts which allow for neuronal communication between different functional regions of the cerebral cortex. These fascicles can be observed and mapped with (DTI), an MRI sequence allowing noninvasive visualization of the microstructural organization of white matter tracts in the brain. Disruption of these fascicles interrupts neural transmission between these regions, resulting in neurological deficits. Techniques designed to avoid fascicular injury have been proposed as a method to avoid damage associated with ICH surgery. Parafascicular surgery is a minimally-invasive technique that, combined with DTI, allows for an atraumatic radial corridor to remove subcortical lesions. This map allows the neurosurgeon to visualize the white matter tracts surrounding the hematoma and to plan the most appropriate and least disruptive surgical tract leading to the hematoma. After obtaining DTI data to create a precise trajectory, the surgeon uses a modified intra-operative computer navigation system to implement a trajectory plan, and introduce a 13 mm circular integrated port under the visualization of an exoscope optics platform. The port has a low coefficient of friction, allowing the surgeon to atraumatically navigate between the fascicles and focally resect the hemorrhage. The combination of these surgical technologies has demonstrated favorable results in excision of brain masses, and has recently been used for evacuation of intracerebral hematomas. Parafascicular surgery with DTI navigation can avoid fascicular damage and collateral injury during ICH evacuation.

1.5 Predictive models for ICH outcome. Several clinical scores have been validated and used to predict mortality and functional outcome after ICH, and have been shown to accurately reflect clinical outcomes, including mortality and functional status. Two of these scores include the modified ICH score and the Essen ICH score. The modified ICH score uses several clinical variables: patient age, presenting National Institutes of Health Stroke Scale (NIHSS) score, hematoma volume and location and presence of intraventricular blood to provide a numerical score that predicts the chances of mortality and of poor functional outcome (defined as ≥2 on the modified Rankin Scale (mRS) at 30 days from presentation. Higher scores are associated with a higher likelihood of poor outcome; scores of 3 are associated with a 70% likelihood of poor outcome, while a score of 5 was associated with mortality rates of 100%. The Essen ICH score was developed to determine the likelihood of functional independence at 100 days from onset. It uses patient age, ICH severity (as measured by NIHSS) and level of consciousness to determine the odds of independent function, measured as a score of 95 or higher on the Barthel index. Patients with low scores (<4) had a 0% chance of achieving functional independence, while 80% of patients with scores >11 were able to live independently at 90 days. Predictive scores have been used in ischemic stroke studies to predict mortality and clinical outcomes. Comparison of outcomes in validated prediction scores is a means to gauge safety and feasibility of intervention.

Hypotheses

This pilot study will evaluate the safety and the clinical outcomes following parafascicular evacuation of ICH in patients selected according to evidence-based criteria.

2.1 Primary objectives: To compare the 30-day and 90-day functional outcomes of patients undergoing parafascicular ICH-evacuation surgery as compared to predicted outcomes using validated ICH prediction scores (the modified ICH score and the Essen ICH score).

2.2 Secondary objectives: To describe and quantify postoperative complications following parafascicular ICH evacuation.

2.3 Hypotheses: We hypothesize that the parafascicular technique will result in equal or reduced mortality, and equal or improved functional outcomes, as compared to ICH predictive scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 presenting with an acute non-traumatic symptomatic supratentorial primary ICH diagnosed by CT
* Severe neurological deficit (National Institutes of Health Stroke Scale (NIHSS) ≥6);
* Symptom onset to surgery < 24 hours (target < 8 hours)
* Glasgow Coma Score greater than or equal to 9
* Hematoma volume <50 millilitres
* Minimal or no ventricular extension (corresponding to 50% or less of each ventricle)

Exclusion Criteria:

* Suspected secondary or traumatic ICH
* Infratentorial ICH
* Isolated intraventricular hemorrhage (IVH)
* Uncorrected coagulopathy
* Significant premorbid disability (mRS >1)
* Hydrocephalus
* Contraindication to safe surgical procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 presenting with an acute non-traumatic symptomatic supratentorial primary ICH diagnosed by CT
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline NIHSS Score at 7 days | 7 days
  Seven days after the procedure, patient NIHSS score(0-42 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of stroke severity.
Change from Baseline Barthel index at 30 days | 30 days
  Thirty days after the procedure, patient Barthel index (0-100 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of functional outcome.
  This assessment will be performed by telephone by an investigator not previously involved in their clinical care. This will be compared to predicted outcome as per modified ICH score.
Change from Baseline Barthel Index at 7 days | 7 days
  Seven days after the procedure, patient Barthel index(0-100 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of change in patient functional status.
Change from Baseline modified Rankin Score at 7 days | 7 days
  Seven days after the procedure, patient mRS score(0-6 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of functional outcome.
Change from Baseline Modified Rankin Score at 30 days | 30 days
  Thirty days after the procedure, patient mRS (0-6 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of functional outcome.
  This assessment will be performed by telephone by an investigator not previously involved in their clinical care. This will be compared to predicted outcome as per modified ICH score.
Mortality at 30 days | 30 days
  Thirty days after the procedure, patients will be contacted for assessment of Barthel index and modified Rankin scale measurement (see other thirty-day outcome measures). At that time, if the patient has died prior to telephone follow-up, the next of kin will be asked for the date and cause of death.
  This assessment will be performed by telephone by an investigator not previously involved in their clinical care. Mortality rate will be compared to predicted outcome as per modified ICH score.
Change from Baseline Barthel index at 90 days | 90 days
  Ninety days after the procedure, patient Barthel index (0-100 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of functional outcome.
  This assessment will be performed by telephone by an investigator not previously involved in their clinical care. This will be compared to predicted outcome as per essen ICH score.
Change from Baseline Modified Rankin Score at 90 days | 90 days
  Ninety days after the procedure, patient mRS (0-6 points)will be measured and compared to baseline (i.e. prior to surgery)as a measure of functional outcome.
  This assessment will be performed by telephone by an investigator not previously involved in their clinical care. This will be compared to predicted outcome as per Essen ICH score.

SECONDARY OUTCOMES:
Presence of post-operative complications between surgery and 30 days | 30 days
  We will collect data on any surgical complications, defined as peri-operative blood loss, thrombotic events, infections, neurological worsening, seizures, metabolic disturbances, and cardiopulmonary events, within 30 days of surgery. We will include data from re-admissions within the first 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Nishihara T, Teraoka A, Morita A, Ueki K, Takai K, Kirino T. A transparent sheath for endoscopic surgery and its application in surgical evacuation of spontaneous intracerebral hematomas. Technical note. J Neurosurg. 2000 Jun;92(6):1053-5. doi: 10.3171/jns.2000.92.6.1053. PMID 10839271
- [Background] McLaughlin N, Prevedello DM, Engh J, Kelly DF, Kassam AB. Endoneurosurgical resection of intraventricular and intraparenchymal lesions using the port technique. World Neurosurg. 2013 Feb;79(2 Suppl):S18.e1-8. doi: 10.1016/j.wneu.2012.02.022. Epub 2012 Feb 10. PMID 22381841